CLINICAL TRIAL: NCT03039790
Title: A Phase 2, Long-Term Immunogenicity Follow-up Trial of Adult and Elderly Subjects Who Have Previously Received an Intramuscular Injection of Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine
Brief Title: Long-Term Immunogenicity of the Norovirus GI.1/GII.4 Bivalent Virus-like Particle (VLP) Vaccine (NoV Vaccine) in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NOR-213; 2016-004288-37 (EudraCT Number); U1111-1189-7907 (Registry Identifier: WHO)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers; Norovirus
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (20):
- NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose (Experimental): Eligible participants who received Hepatitis A vaccine, intramuscular (IM), on Day 1, followed by norovirus bivalent virus like particle (VLP) vaccine (15 µg of GI.1 norovirus virus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 50 µg monophosphoryl lipid A (MLP) and 500 µg aluminium hydroxide, IM on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MPL and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MPL and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 15 µg MPL and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose (Experimental): Eligible NOR-107 participants who had received IM hepatitis A vaccine on Day 1, followed by IM norovirus bivalent vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MPL and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MPL and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 150 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose (Experimental): Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose (Experimental): Eligible NOR-107 participants who had received Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 1 and Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose (Experimental): Eligible NOR-107 participants who had received Norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 150 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 1 and Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose (Experimental): Eligible NOR-107 participants who had received Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminium hydroxide, IM, on Day 1 and Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose (Experimental): Eligible NOR-210 participants who had received Norovirus GI.1/GII.4 bivalent VLP vaccine NoV Vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP, adjuvanted with 500 µg aluminium hydroxide), IM injection, once on Day 1 were enrolled at 2nd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose (Experimental): Eligible NOR-204 participants who had received Norovirus bivalent placebo-matching vaccine, intramuscularly (IM), on Day 1, followed by norovirus (NoV) [15 μg of GI.1 and 50 μg of GII.4 bivalent virus-like particle (VLP)] adjuvanted with 500 µg aluminium hydroxide and 15 μg of monophosphoryl lipid A (MPL) (Composition B), on Day 29 were enrolled at 2nd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 yrs) (Experimental): Eligible NOR-204 participants of age 60-94 years who had received Norovirus bivalent placebo-matching vaccine, IM, on Day 1, followed by norovirus (NoV) [15 μg of GI.1 and 50 μg of GII.4 bivalent virus-like particle (VLP)] adjuvanted with 500 µg aluminium hydroxide (Composition A), on Day 29 were enrolled at 2nd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 yrs) (Experimental): Eligible NOR-204 participants of age 18-49 years who had received Norovirus bivalent placebo-matching vaccine, IM, on Day 1, followed by norovirus (NoV) [15 μg of GI.1 and 50 μg of GII.4 bivalent virus-like particle (VLP)] adjuvanted with 500 µg aluminium hydroxide (Composition A), on Day 29 were enrolled at 2nd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose (Experimental): Eligible NOR-204 participants who had received Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide and 15 μg of MPL (Composition B), IM, on Day 1 and Day 29 were enrolled at 2nd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine
- NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose (Experimental): Eligible NOR-204 participants who had received Norovirus bivalent placebo-matching vaccine (15 μg of GI.1 50 μg of GII.4 bivalent VLP) adjuvanted with 500 µg aluminium hydroxide (Composition A) IM, on Day 1 and Day 29 were enrolled at 2nd year post-primary vaccination in NOR-213 study.
  Interventions: Biological: NoV Vaccine

INTERVENTIONS:
Biological: NoV Vaccine — NoV vaccine injection administered.

SUMMARY:
The purpose of this study is to evaluate descriptively the long-term immunogenicity of at least 1 NoV vaccine administration.

DETAILED DESCRIPTION:
Results prepared and posted by Takeda on behalf of Hillevax, the IND holder.

The drug being tested in this study is called NoV vaccine. NoV vaccine is being tested for protection against acute gastroenteritis (AGE) due to norovirus.

The study will enroll maximum of approximately 575 participants. Participants who previously received NoV vaccine in studies NOR-107, NOR-210 and NOR-204 will be enrolled. Participants from study NOR-107 will enter the study at the time of their 3rd year post-primary vaccination, and from studies NOR-210 and NOR-204, at their 2nd year post-primary vaccination. The duration of participation in the study will be different for each participant.

This multi-center trial will be conducted in Belgium and the United States. The overall time to participate in this study is maximum 5 years after primary NoV vaccination. Participants will have a maximum of 4 visits over 3 years

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants who previously received at least 1 dose of NoV vaccine in trials NOR-107 (NCT02038907), NOR-210 (NCT02475278) and NOR-204 (NCT02661490), have baseline and post-vaccination data, and completed the primary vaccination trial protocol as initially described.

Exclusion Criteria:

1. Participation in any clinical trial is allowed, on condition that no investigational product is administered within 30 days prior to blood sampling.
2. In the opinion of the investigator, the participant is not medically eligible to provide blood specimens.
3. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (11):
- United States (9):
  - Simon-Williamson Clinic/Synexus Clinical Research US, Inc, Birmingham, Alabama
  - Synexus Clinical Research US, Inc./Fountain Hills Family Practice, P.C., Fountain Hills, Arizona
  - Synexus Clinical Research US, Inc/Southwest Family Medicine, Littleton, Colorado
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - St. Louis University, School of Medicine, St Louis, Missouri
  - Regional Clinical Research Inc., Endwell, New York
  - University of Rochester, Rochester, New York
  - Benchmark Research Austin, Austin, Texas
- Belgium (2):
  - Universiteit Antwerpen, Antwerp
  - Universitair Ziekenhuis Gent, Ghent

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Groups:
- NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose: Eligible NOR-107 participants who had received Hepatitis A vaccine, intramuscular (IM), on Day 1, followed by norovirus bivalent virus like particle (VLP) vaccine (15 µg of GI.1 norovirus virus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 50 µg monophosphoryl lipid A (MPL) and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
Period: Overall Study
Arm/Group | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose
Started | 25 | 19 | 27 | 27 | 23 | 27 | 25 | 28 | 22 | 28 | 21 | 25 | 24 | 24 | 24 | 29 | 39 | 14 | 35 | 42
Per Protocol Set (PPS) (PPS included all participants in the FAS who had no major or critical protocol violations that potentially confound the primary endpoint.) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 24 | 29 | 39 | 14 | 35 | 42
Completed | 21 | 19 | 26 | 25 | 23 | 26 | 24 | 27 | 22 | 26 | 20 | 25 | 21 | 24 | 20 | 22 | 29 | 12 | 29 | 34
Not Completed | 4 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 3 | 0 | 4 | 7 | 10 | 2 | 6 | 8
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 2 | 2 | 1 | 3
Not completed — Withdrawal of Consent | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 5 | 3 | 0 | 2 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0
Not completed — Reason, not Specified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants with data from at least 1 follow-up time point.
Groups:
- NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose: Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
- NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose: Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
- NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose: Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
- NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose: Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 150 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
- NOR-107: GI.1/GII.4 (15/150/167) μg,1-Dose: Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
- Total: Total of all reporting groups
Arm/Group | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose | NOR-107: GI.1/GII.4 (15/150/167) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose | Total
Number analyzed (Participants) | 25 | 19 | 27 | 27 | 23 | 27 | 25 | 28 | 22 | 28 | 21 | 25 | 24 | 24 | 24 | 29 | 39 | 14 | 35 | 42 | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (14.24) | 47.9 (14.60) | 46.8 (13.39) | 47.5 (13.96) | 48.0 (13.49) | 48.0 (13.13) | 45.4 (13.63) | 46.8 (13.59) | 45.5 (13.23) | 44.0 (15.20) | 41.9 (16.17) | 42.6 (13.33) | 47.3 (13.98) | 46.3 (15.17) | 35.0 (9.44) | 73.6 (8.50) | 77.2 (9.48) | 35.6 (7.27) | 76.9 (9.94) | 76.1 (8.41) | 53.6 (18.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 19 | 20 | 14 | 21 | 12 | 14 | 16 | 21 | 12 | 15 | 18 | 16 | 10 | 20 | 19 | 7 | 18 | 23 | 324
  Male | 9 | 6 | 8 | 7 | 9 | 6 | 13 | 14 | 6 | 7 | 9 | 10 | 6 | 8 | 14 | 9 | 20 | 7 | 17 | 19 | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 1 | 3 | 3 | 15
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 28 | 37 | 13 | 32 | 39 | 168
  Unknown or Not Reported | 25 | 19 | 27 | 27 | 23 | 27 | 25 | 28 | 22 | 28 | 21 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 345
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 1 | 0 | 3 | 12
  White | 25 | 19 | 27 | 26 | 23 | 26 | 25 | 28 | 22 | 27 | 21 | 25 | 24 | 24 | 16 | 28 | 38 | 12 | 35 | 39 | 510
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 25 | 19 | 27 | 27 | 23 | 27 | 25 | 28 | 22 | 28 | 21 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 345
  United States | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 29 | 39 | 14 | 35 | 42 | 183

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Blocking Titers 50 Percent (%) (GMBT50) of Anti-norovirus GI.1 VLP Antibodies as Measured by Histo-Blood Group Antigen HBGA Blocking Assay
Description: GMBT50 of anti-norovirus GI. VLP antibody titers as measured by the histo-blood group antigen (HBGA) blocking assay. Data reported for up to Year 5 was collected at Baseline (NOR-107, NOR-210, NOR-204) , at Days 28 (NOR-107), 29 (NOR-204 and NOR-210), Day 36 (NOR-204), Day 56 (NOR-107) and Day 57 (NOR-204), Day 208 (NOR-107) and Day 211 (NOR-204), Year 2 (NOR-204 and NOR-210) Years 3, 4 and 5 (NOR-107, NOR-210, NOR-204)
Time Frame: Baseline up to Year 2 post-primary vaccination of initial study NOR-107, NOR-210 NOR-204 and up to Year 5 of this extension study
Population: Per Protocol Set (PPS) included all participants in the FAS who had no major or critical protocol violations that potentially confound the primary endpoint. Number analyzed is the number of participants with data available for analysis at specific timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose
Number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 24 | 29 | 39 | 14 | 35 | 42
titer
  Baseline | 27.4 [17.5 to 42.9] | 18.3 [13.4 to 24.9] | 26.3 [17.4 to 39.6] | 24.6 [15.5 to 38.9] | 19.0 [15.5 to 23.2] | 23.9 [17.2 to 33.2] | 35.1 [21.7 to 56.9] | 24.3 [16.5 to 35.8] | 26.1 [16.8 to 40.5] | 23.9 [17.5 to 32.7] | 33.4 [19.4 to 57.6] | 23.1 [16.4 to 32.6] | 22.9 [15.9 to 32.9] | 21.3 [15.4 to 29.3] | 19.0 [14.1 to 25.6] | 20.8 [16.4 to 26.3] | 28.9 [20.7 to 40.5] | 18.7 [13.0 to 26.9] | 23.9 [18.5 to 30.8] | 26.4 [19.4 to 36.1]
  Days 28: number analyzed (Participants) | 25 | 19 | 26 | 26 | 23 | 27 | 25 | 28 | 21 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Days 28 | 27.7 [18.2 to 42.2] | 18.1 [13.2 to 24.8] | 23.8 [16.4 to 34.5] | 24.0 [15.4 to 37.3] | 17.4 [14.5 to 20.9] | 21.9 [16.1 to 29.9] | 29.9 [20.2 to 44.2] | 24.9 [17.2 to 36.1] | 27.3 [17.2 to 43.4] | 25.8 [18.3 to 36.3] | 34.9 [20.8 to 58.5] | 382.6 [200.9 to 728.5] | 338.0 [196.7 to 580.7] | 449.4 [270.5 to 746.5] |  |  |  |  |  |
  Days 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 29 | 39 | 14 | 35 | 42
  Days 29 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 212.5 [129.9 to 347.5] | 21.3 [16.9 to 26.9] | 28.7 [20.6 to 40.0] | 19.9 [13.5 to 29.2] | 342.5 [206.3 to 568.5] | 329.2 [213.3 to 508.2]
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 36 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 263.3 [143.3 to 483.9] | 213.4 [117.2 to 388.5] | 155.3 [51.5 to 468.2] | 406.4 [274.6 to 601.4] | 307.2 [206.1 to 458.0]
  Day 56: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 56 | 309.7 [168.7 to 568.4] | 256.9 [136.3 to 484.0] | 380.9 [227.0 to 639.2] | 255.4 [132.3 to 493.1] | 252.9 [136.7 to 468.1] | 329.2 [192.9 to 561.9] | 369.5 [221.0 to 617.8] | 350.4 [194.5 to 631.2] | 527.0 [264.1 to 1051.5] | 274.3 [171.6 to 438.4] | 315.8 [154.5 to 645.2] | 435.9 [288.8 to 658.0] | 427.6 [300.0 to 609.6] | 377.4 [251.6 to 566.0] |  |  |  |  |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 57 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 228.9 [136.4 to 384.1] | 223.0 [133.9 to 371.5] | 105.1 [40.9 to 270.5] | 362.5 [255.9 to 513.5] | 304.3 [215.6 to 429.7]
  Day 208: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 208 | 143.5 [84.7 to 243.2] | 109.1 [62.9 to 189.1] | 154.8 [95.7 to 250.4] | 125.6 [74.9 to 210.8] | 86.4 [50.5 to 148.1] | 137.9 [93.7 to 202.8] | 168.9 [109.1 to 261.5] | 175.4 [111.6 to 275.6] | 214.1 [120.7 to 379.6] | 125.3 [83.7 to 187.6] | 115.3 [61.5 to 216.0] | 208.7 [134.0 to 324.9] | 201.5 [141.3 to 287.4] | 185.6 [126.9 to 271.6] |  |  |  |  |  |
  Day 211: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 211 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 115.9 [72.1 to 186.4] | 96.5 [62.6 to 148.7] | 43.4 [20.1 to 93.9] | 132.9 [89.2 to 198.0] | 126.6 [85.6 to 187.2]
  Year 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 26 | 37 | 14 | 32 | 34
  Year 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 48.8 [31.2 to 76.4] | 46.3 [30.7 to 69.8] | 63.6 [39.6 to 102.1] | 38.9 [16.7 to 90.6] | 58.9 [39.8 to 87.2] | 83.4 [58.2 to 119.3]
  Year 3: number analyzed (Participants) | 24 | 19 | 27 | 26 | 23 | 26 | 25 | 28 | 22 | 27 | 19 | 25 | 24 | 24 | 21 | 24 | 35 | 13 | 29 | 37
  Year 3 | 79.6 [48.9 to 129.7] | 53.7 [32.8 to 88.0] | 77.2 [49.1 to 121.3] | 72.4 [44.0 to 119.1] | 51.5 [33.1 to 80.1] | 55.5 [35.4 to 86.8] | 98.0 [65.1 to 147.5] | 90.2 [60.1 to 135.5] | 102.2 [56.4 to 185.0] | 61.8 [40.5 to 94.3] | 67.2 [34.5 to 131.1] | 90.5 [55.4 to 147.6] | 84.9 [53.1 to 135.6] | 85.7 [55.9 to 131.4] | 48.2 [29.0 to 80.1] | 48.8 [30.3 to 78.8] | 60.7 [37.2 to 98.9] | 34.0 [16.6 to 69.9] | 72.5 [47.3 to 111.2] | 76.1 [51.0 to 113.6]
  Year 4: number analyzed (Participants) | 23 | 19 | 26 | 26 | 23 | 26 | 23 | 28 | 22 | 28 | 19 | 25 | 23 | 24 | 20 | 18 | 22 | 11 | 20 | 27
  Year 4 | 70.5 [38.0 to 130.9] | 47.5 [27.3 to 82.7] | 68.6 [38.6 to 122.0] | 54.0 [30.4 to 96.1] | 54.8 [30.2 to 99.7] | 49.3 [31.5 to 77.2] | 84.9 [49.6 to 145.2] | 67.3 [41.1 to 109.9] | 78.2 [41.9 to 146.1] | 45.5 [30.0 to 68.9] | 61.2 [30.9 to 121.0] | 85.8 [57.9 to 127.0] | 65.1 [39.0 to 108.8] | 67.2 [42.9 to 105.2] | 63.8 [35.0 to 116.2] | 28.6 [17.3 to 47.2] | 45.9 [25.0 to 84.3] | 28.3 [14.2 to 56.2] | 76.1 [45.6 to 127.2] | 57.1 [34.5 to 94.3]
  Year 5: number analyzed (Participants) | 21 | 19 | 26 | 24 | 23 | 26 | 24 | 27 | 22 | 25 | 19 | 24 | 21 | 24 | 19 | 8 | 13 | 10 | 10 | 16
  Year 5 | 71.0 [37.8 to 133.6] | 42.5 [25.0 to 72.4] | 80.5 [45.0 to 144.0] | 54.4 [30.8 to 96.2] | 50.5 [28.7 to 89.1] | 54.5 [31.0 to 96.0] | 77.2 [48.4 to 123.1] | 82.2 [49.0 to 137.7] | 80.9 [43.3 to 151.1] | 54.1 [32.6 to 89.7] | 62.0 [32.5 to 118.5] | 82.1 [50.9 to 132.4] | 69.1 [42.3 to 112.6] | 74.9 [49.1 to 114.2] | 52.8 [28.6 to 97.4] | 34.7 [15.8 to 76.1] | 41.9 [21.8 to 80.3] | 31.9 [14.6 to 69.6] | 59.8 [29.0 to 123.2] | 65.5 [37.9 to 113.1]

2. Primary Outcome: Geometric Mean Blocking Titer (GMBT50) of Anti-norovirus GII.4 VLP Antibodies as Measured by HBGA Blocking Assay
Description: GMBT50 of anti-norovirus GII.4 VLP antibody titers as measured by the HBGA blocking assay. Data reported for up to Year 5 was collected at Baseline (NOR-107, NOR-210, NOR-204), at Days 28 (NOR-107), 29 (NOR-204 and NOR-210), Day 36 (NOR-204), Day 56 (NOR-107) and Day 57 (NOR-204), Day 208 (NOR-107) and Day 211 (NOR-204), Year 2 (NOR-204 and NOR-210) Years 3 4 and 5 (NOR-107,NOR-210, NOR-204) .
Time Frame: as for outcome 1
Population: PPS included all participants in the FAS who had no major or critical protocol violations that potentially confound the primary endpoint. Number analyzed is the number of participants with data available for analysis at specific timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose: Eligible participants who received IM hepatitis A vaccine on Day 1, followed by IM norovirus bivalent vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MLP and 500 µg aluminium hydroxide, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose: Eligible NOR-107 participants who had received IM hepatitis A vaccine on Day 1, followed by IM norovirus bivalent vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MPL and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
- NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose: Eligible NOR-107 participants who had received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MPL and 500 µg aluminium hydroxide, on Day 28 were enrolled at 3rd year post-primary vaccination in NOR-213 study.
- NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 150 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (15/15/167) μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (50/50/500) μg,2-Dose: Eligible participants who received Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 1 and Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose: Eligible participants who received Norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 150 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 1 and Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose: Eligible participants who received Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminium hydroxide, IM, on Day 1 and Day 28in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose: Eligible participants who received Norovirus GI.1/GII.4 bivalent VLP vaccine NoV Vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP, adjuvanted with 500 µg aluminium hydroxide), IM injection, once on Day 1 in previous study NOR-210 were enrolled at 2nd year post-primary vaccination in this study.
- NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose: Eligible participants ≥ 60 years of age, received 1-dose regimen: Norovirus bivalent placebo-matching vaccine, intramuscularly (IM), on Day 1, followed by norovirus (NoV) GI.1 (15 μg)/GII.4 (50 μg) bivalent virus-like particle (VLP) vaccine (Formulation A), IM, on Day 29 in previous study NOR-204 were enrolled at 2nd year post-primary vaccination in this study.
- NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs): Eligible participants 60-94 years of age, received 1-dose regimen: Norovirus bivalent placebo-matching vaccine, IM on Day 1, followed by norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine with 15 μg monophosphoryl lipid A (MPL) (Formulation B), IM, on Day 29 in previous study NOR-204 were enrolled at 2nd year post-primary vaccination in this study.
- NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs): Eligible participants 18 to 49 years of age, received 1-dose regimen: Norovirus bivalent placebo-matching vaccine, IM, on Day 1, followed by norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine (Formulation A), IM, on Day 29 in previous study NOR-204 were enrolled at 2nd year post-primary vaccination in this study.
- NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose: Eligible participants ≥ 60 years of age, received 2-dose regimen: Norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine with 15 μg MPL (Formulation B), IM, on Days 1 and 29 in previous study NOR-204 were enrolled at 2nd year post-primary vaccination in this study.
- NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose: Eligible participants ≥ 60 years of age, received 2-dose regimen: Norovirus bivalent placebo-matching vaccine, IM, on Day 1, followed by norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine (Formulation A), IM, on Day 29 in previous study NOR-204 were enrolled at 2nd year post-primary vaccination in this study.
Arm/Group | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/167) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,2-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose
Number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 24 | 29 | 39 | 14 | 35 | 42
titer
  Baseline | 74.8 [38.1 to 147.0] | 77.4 [41.9 to 142.8] | 116.8 [65.9 to 207.2] | 72.1 [41.6 to 125.1] | 54.6 [30.7 to 97.3] | 104.2 [60.4 to 179.8] | 77.5 [42.5 to 141.6] | 86.3 [47.9 to 155.3] | 97.1 [55.8 to 169.0] | 106.1 [66.7 to 168.8] | 124.3 [69.0 to 223.9] | 65.8 [39.6 to 109.1] | 97.2 [53.8 to 175.9] | 127.3 [70.2 to 231.0] | 42.7 [25.6 to 71.1] | 140.5 [78.5 to 251.6] | 71.8 [45.7 to 113.0] | 97.5 [40.3 to 235.8] | 104.9 [64.2 to 171.5] | 111.0 [72.0 to 171.1]
  Day 28: number analyzed (Participants) | 25 | 19 | 26 | 26 | 23 | 27 | 25 | 28 | 21 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 28 | 80.7 [42.3 to 153.9] | 67.2 [35.2 to 128.0] | 128.0 [73.3 to 223.7] | 71.3 [42.2 to 120.7] | 64.9 [36.6 to 115.3] | 101.3 [57.1 to 179.6] | 69.7 [40.2 to 120.9] | 95.2 [49.6 to 182.6] | 84.1 [46.7 to 151.3] | 129.9 [83.4 to 202.4] | 112.4 [63.0 to 200.5] | 607.7 [379.2 to 974.0] | 668.3 [397.3 to 1124.0] | 893.6 [578.4 to 1380.5] |  |  |  |  |  |
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 29 | 39 | 14 | 35 | 42
  Day 29 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 665.9 [408.2 to 1086.2] | 118.3 [66.7 to 210.0] | 63.5 [41.0 to 98.4] | 83.2 [34.3 to 201.9] | 1134.4 [784.6 to 1640.1] | 824.2 [493.4 to 1376.8]
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 36 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 920.9 [521.8 to 1625.4] | 518.7 [273.0 to 985.2] | 1037.4 [448.1 to 2401.9] | 1016.2 [719.4 to 1435.4] | 766.8 [483.1 to 1216.9]
  Day 56: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 56 | 367.9 [214.8 to 630.3] | 755.9 [425.6 to 1342.6] | 425.1 [298.8 to 604.8] | 277.9 [178.2 to 433.4] | 584.7 [367.5 to 930.1] | 593.4 [436.2 to 807.2] | 201.9 [110.6 to 368.4] | 810.0 [507.4 to 1293.2] | 328.5 [173.8 to 620.8] | 886.3 [562.3 to 1397.0] | 746.6 [456.8 to 1220.3] | 458.4 [290.9 to 722.3] | 575.5 [358.1 to 924.8] | 594.2 [369.2 to 956.2] |  |  |  |  |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 57 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1133.2 [682.7 to 1881.0] | 471.8 [285.2 to 780.5] | 663.8 [304.5 to 1447.1] | 740.2 [549.0 to 998.0] | 589.1 [359.7 to 964.6]
  Day 208: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 208 | 216.4 [132.8 to 352.6] | 290.1 [182.7 to 460.7] | 231.4 [152.0 to 352.4] | 176.2 [116.1 to 267.4] | 215.9 [132.1 to 353.1] | 247.4 [166.6 to 367.3] | 150.4 [87.4 to 258.6] | 333.2 [217.9 to 509.4] | 173.0 [94.8 to 315.8] | 352.9 [242.4 to 513.8] | 274.9 [151.4 to 499.2] | 277.2 [186.5 to 412.0] | 342.5 [233.2 to 503.1] | 308.7 [198.5 to 480.0] |  |  |  |  |  |
  Day 211: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 211 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 417.6 [252.8 to 689.6] | 195.2 [120.2 to 316.8] | 274.7 [135.3 to 557.8] | 374.7 [262.6 to 534.6] | 265.3 [157.4 to 447.2]
  Year 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 26 | 37 | 10 | 32 | 35
  Year 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 105.2 [58.7 to 188.3] | 223.2 [120.7 to 412.9] | 122.5 [74.8 to 200.5] | 250.5 [80.8 to 776.7] | 220.9 [137.2 to 355.7] | 243.0 [149.6 to 394.7]
  Year 3: number analyzed (Participants) | 24 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 27 | 19 | 25 | 24 | 24 | 21 | 24 | 35 | 13 | 29 | 37
  Year 3 | 122.7 [65.7 to 229.2] | 177.1 [96.8 to 323.9] | 117.9 [69.6 to 199.7] | 104.0 [60.2 to 179.6] | 80.5 [45.4 to 142.9] | 125.9 [74.7 to 212.3] | 121.2 [71.1 to 206.7] | 164.1 [97.7 to 275.5] | 125.3 [67.9 to 230.9] | 167.0 [111.3 to 250.4] | 142.2 [76.9 to 263.1] | 149.2 [83.1 to 267.9] | 144.7 [83.1 to 251.7] | 173.8 [104.6 to 288.8] | 87.5 [43.9 to 174.5] | 172.0 [100.1 to 295.5] | 94.9 [59.4 to 151.3] | 133.8 [56.2 to 318.9] | 153.3 [100.1 to 234.8] | 162.4 [102.5 to 257.3]
  Year 4: number analyzed (Participants) | 23 | 19 | 26 | 26 | 23 | 26 | 23 | 28 | 22 | 28 | 19 | 25 | 23 | 24 | 20 | 18 | 22 | 11 | 20 | 27
  Year 4 | 85.7 [46.7 to 157.1] | 122.8 [67.4 to 223.6] | 90.8 [54.4 to 151.3] | 79.5 [48.3 to 130.8] | 61.7 [35.7 to 106.5] | 106.7 [64.7 to 176.1] | 108.6 [62.0 to 190.3] | 131.2 [81.9 to 210.2] | 101.9 [60.1 to 172.7] | 113.9 [73.3 to 177.1] | 130.1 [70.0 to 241.9] | 98.1 [55.0 to 175.1] | 104.4 [58.4 to 186.5] | 120.3 [72.6 to 199.3] | 84.1 [44.2 to 160.3] | 116.0 [54.0 to 249.4] | 80.9 [42.1 to 155.4] | 131.1 [57.6 to 298.6] | 241.9 [140.2 to 417.5] | 136.7 [75.7 to 246.9]
  Year 5: number analyzed (Participants) | 21 | 19 | 26 | 24 | 23 | 26 | 24 | 27 | 22 | 25 | 19 | 24 | 21 | 24 | 19 | 8 | 14 | 10 | 10 | 17
  Year 5 | 101.1 [52.5 to 194.6] | 138.3 [80.8 to 236.9] | 124.4 [78.5 to 197.0] | 91.2 [51.2 to 162.3] | 71.3 [40.0 to 126.9] | 103.2 [60.6 to 175.8] | 94.3 [54.4 to 163.2] | 144.9 [82.9 to 253.1] | 105.1 [57.8 to 191.1] | 147.2 [92.4 to 234.4] | 118.0 [66.8 to 208.6] | 118.3 [71.4 to 195.8] | 115.7 [57.7 to 232.0] | 132.0 [79.7 to 218.5] | 94.2 [49.1 to 180.7] | 123.4 [26.5 to 574.3] | 66.8 [32.2 to 138.6] | 107.4 [43.5 to 265.1] | 202.2 [110.2 to 370.9] | 187.3 [105.6 to 332.4]

3. Secondary Outcome: Geometric Mean Titers (GMT) of Anti-norovirus GI.1 VLP Antibodies as Measured by Total Immunoglobulin (Pan-Ig) Enzyme-linked Immunosorbent Assay (ELISA)
Description: GMT of anti-norovirus GI.1 VLP antibody titers as measured by total immunoglobulin (pan-Ig) enzyme-linked immunoassay (ELISA). Data reported for up to Year 5 was collected at Baseline (NOR-107, NOR-210, NOR-204), at Days 28 (NOR-107), 29 (NOR-204 and NOR-210), Day 36 (NOR-204), Day 56 (NOR-107) and Day 57 (NOR-204), Day 208 (NOR-107) and Day 211 (NOR-204), Year 2 (NOR-204 and NOR-210) Years 3, 4 and 5(NOR-107,NOR-210, NOR-204).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MLP and 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 15 µg MLP and 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 15 µg MLP and 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 167 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
- NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose: Eligible participants who received Norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminium hydroxide, IM, on Day 1 and Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
Arm/Group | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose
Number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 24 | 29 | 39 | 14 | 35 | 42
titer
  Baseline | 1030.5 [543.6 to 1953.7] | 689.8 [295.3 to 1611.4] | 646.2 [354.3 to 1178.4] | 620.9 [326.7 to 1180.1] | 547.4 [334.5 to 895.6] | 539.6 [293.3 to 992.5] | 1089.2 [599.9 to 1977.6] | 856.1 [471.5 to 1554.3] | 749.7 [406.6 to 1382.5] | 770.6 [413.5 to 1436.2] | 925.3 [366.0 to 2339.3] | 777.3 [413.1 to 1462.8] | 908.6 [501.0 to 1647.8] | 640.4 [378.5 to 1083.5] | 160.1 [78.6 to 326.1] | 671.5 [432.5 to 1042.4] | 769.8 [559.5 to 1059.0] | 493.1 [170.7 to 1424.8] | 683.8 [460.7 to 1014.9] | 851.8 [534.3 to 1357.9]
  Day 28: number analyzed (Participants) | 25 | 19 | 26 | 26 | 23 | 27 | 25 | 28 | 21 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 28 | 975.2 [508.7 to 1869.6] | 649.3 [285.2 to 1478.2] | 544.9 [297.5 to 998.3] | 648.7 [324.3 to 1297.5] | 475.4 [284.8 to 793.4] | 535.4 [287.5 to 997.1] | 1086.1 [613.7 to 1922.0] | 839.1 [469.7 to 1499.0] | 729.3 [380.1 to 1399.5] | 731.0 [382.7 to 1396.2] | 932.8 [402.0 to 2164.8] | 16822.8 [11052.9 to 25604.9] | 21215.2 [15921.0 to 28269.9] | 14102.7 [9666.5 to 20574.8] |  |  |  |  |  |
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 29 | 39 | 14 | 35 | 42
  Day 29 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 10798.6 [7482.3 to 15584.8] | 630.6 [407.9 to 974.8] | 734.8 [544.2 to 992.1] | 694.7 [249.8 to 1931.4] | 10862.2 [8363.3 to 14107.7] | 8286.7 [6204.3 to 11068.0]
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 36 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 6915.9 [4770.3 to 10026.5] | 3909.4 [2555.3 to 5981.0] | 7407.6 [3545.0 to 15479.0] | 10851.2 [8549.3 to 13772.9] | 8143.0 [6132.6 to 10812.4]
  Day 56: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 56 | 15032.5 [10033.4 to 22522.2] | 12246.2 [7488.7 to 20025.9] | 16739.1 [11460.0 to 24450.0] | 13673.2 [8411.3 to 22226.9] | 12847.2 [9036.9 to 18264.2] | 18464.0 [14207.7 to 23995.3] | 15242.3 [11298.2 to 20563.2] | 15071.0 [9104.8 to 24946.5] | 25738.6 [16696.8 to 39676.9] | 14709.3 [10110.9 to 21399.2] | 12428.4 [6942.7 to 22248.5] | 14302.9 [10081.6 to 20291.8] | 18086.8 [13594.7 to 24063.2] | 11282.4 [8142.8 to 15632.5] |  |  |  |  |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 57 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 10684.3 [8532.4 to 13378.9] | 5646.8 [4043.4 to 7886.1] | 7944.8 [4570.2 to 13811.2] | 9388.2 [7285.3 to 12098.2] | 7316.3 [5685.6 to 9414.7]
  Day 208: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 208 | 6015.9 [4271.9 to 8471.9] | 4784.5 [3114.9 to 7349.0] | 6231.0 [4321.0 to 8985.3] | 5675.5 [3783.7 to 8513.4] | 4212.3 [3065.0 to 5789.1] | 4997.4 [3748.7 to 6662.0] | 5577.8 [4072.7 to 7639.2] | 6686.7 [4766.4 to 9380.5] | 7761.2 [5226.5 to 11525.1] | 5274.3 [3746.7 to 7424.6] | 4978.7 [3275.4 to 7567.6] | 7082.7 [5051.7 to 9930.2] | 7469.9 [5874.5 to 9498.6] | 5355.9 [4082.7 to 7026.2] |  |  |  |  |  |
  Day 211: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 211 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 5970.0 [4586.1 to 7771.7] | 4137.3 [3176.2 to 5389.2] | 3745.8 [1975.8 to 7101.5] | 5320.5 [4169.4 to 6789.4] | 5020.4 [3878.5 to 6498.6]
  Year 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 26 | 37 | 10 | 32 | 35
  Year 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1662.0 [1203.1 to 2296.0] | 1804.4 [1405.6 to 2316.4] | 1477.4 [1016.3 to 2147.7] | 1672.4 [656.0 to 4263.7] | 1770.6 [1310.4 to 2392.3] | 1635.0 [1194.2 to 2238.4]
  Year 3: number analyzed (Participants) | 24 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 27 | 19 | 25 | 24 | 24 | 21 | 24 | 35 | 13 | 29 | 37
  Year 3 | 2229.0 [1481.3 to 3354.1] | 1493.3 [987.8 to 2257.6] | 2058.7 [1538.0 to 2755.7] | 2227.0 [1581.4 to 3136.2] | 1465.7 [1056.7 to 2032.8] | 1568.0 [1188.6 to 2068.5] | 2156.1 [1527.7 to 3042.9] | 1913.2 [1386.8 to 2639.4] | 2063.1 [1370.8 to 3105.0] | 1702.4 [1165.5 to 2486.6] | 1579.5 [977.5 to 2552.2] | 2422.7 [1732.0 to 3388.9] | 2914.8 [2270.4 to 3742.1] | 2077.8 [1523.3 to 2834.1] | 1500.9 [1031.3 to 2184.2] | 2006.4 [1373.3 to 2931.3] | 1932.8 [1245.7 to 2998.7] | 1254.9 [701.7 to 2244.2] | 1670.1 [1258.5 to 2216.4] | 1700.5 [1224.7 to 2361.3]
  Year 4: number analyzed (Participants) | 23 | 19 | 26 | 26 | 23 | 26 | 23 | 28 | 22 | 28 | 19 | 25 | 23 | 24 | 20 | 18 | 22 | 11 | 20 | 27
  Year 4 | 2095.5 [1272.0 to 3452.2] | 1727.7 [1016.1 to 2937.8] | 2541.1 [1618.3 to 3990.1] | 1958.2 [1363.0 to 2813.3] | 1802.9 [1185.9 to 2740.8] | 1565.5 [1181.0 to 2075.1] | 2934.1 [1993.0 to 4319.7] | 2107.0 [1384.3 to 3207.0] | 1965.0 [1287.9 to 2997.9] | 1679.0 [1208.0 to 2333.5] | 2025.2 [1254.9 to 3268.3] | 2335.8 [1724.4 to 3163.8] | 2635.7 [1936.2 to 3587.9] | 2016.6 [1500.0 to 2711.1] | 1627.4 [1127.0 to 2350.1] | 1512.1 [1032.5 to 2214.6] | 1441.7 [926.9 to 2242.4] | 1238.3 [841.5 to 1822.1] | 1585.6 [1101.6 to 2282.3] | 1392.4 [917.6 to 2112.9]
  Year 5: number analyzed (Participants) | 21 | 19 | 26 | 24 | 23 | 26 | 24 | 27 | 22 | 25 | 19 | 24 | 21 | 24 | 19 | 8 | 15 | 10 | 10 | 16
  Year 5 | 1732.3 [1133.8 to 2646.8] | 1563.6 [957.9 to 2552.6] | 2345.8 [1566.6 to 3512.7] | 2009.8 [1396.6 to 2892.2] | 1664.8 [1100.7 to 2518.1] | 1781.2 [1102.5 to 2877.7] | 2116.5 [1597.7 to 2803.7] | 2270.3 [1536.1 to 3355.5] | 2181.9 [1360.4 to 3499.2] | 1811.9 [1173.5 to 2797.8] | 1434.9 [956.9 to 2151.6] | 2036.9 [1475.0 to 2812.9] | 2405.4 [1763.1 to 3281.8] | 1817.7 [1256.1 to 2630.5] | 1803.8 [1205.4 to 2699.1] | 1937.4 [1141.5 to 3288.2] | 1255.5 [709.1 to 2223.1] | 1048.6 [566.7 to 1940.4] | 2060.5 [1422.7 to 2984.3] | 1687.2 [1031.7 to 2759.3]

4. Secondary Outcome: Geometric Mean Titers (GMT) of Anti-norovirus GII.4 VLP Antibodies as Measured by Pan-Ig ELISA
Description: GMT of anti-norovirus GII.4 VLP antibody titers as measured by pan-Ig ELISA. Data reported for up to Year 5 was collected at Baseline (NOR-107,NOR-210, NOR-204), at Days 28 (NOR-107), 29 (NOR-204 and NOR-210), Day 36 (NOR-204), Day 56 (NOR-107) and Day 57 (NOR-204), Day 208 (NOR-107) and Day 211 (NOR-204), Year 2 (NOR-204 and NOR-210) Years 3, 4 and 5 (NOR-107,NOR-210, NOR-204).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose
Number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 24 | 29 | 39 | 14 | 35 | 42
titer
  Baseline | 1209.8 [617.2 to 2371.5] | 1248.3 [665.1 to 2343.0] | 1423.3 [799.5 to 2533.7] | 954.0 [530.1 to 1716.8] | 838.8 [507.6 to 1386.1] | 1239.7 [705.8 to 2177.4] | 1373.7 [792.4 to 2381.6] | 1179.5 [677.5 to 2053.4] | 1133.9 [648.4 to 1982.8] | 1442.1 [864.3 to 2406.1] | 2069.2 [1362.0 to 3143.7] | 1078.9 [678.4 to 1715.6] | 1308.9 [779.3 to 2198.4] | 1598.5 [952.6 to 2682.3] | 93.1 [58.8 to 147.3] | 1213.2 [658.2 to 2236.1] | 826.1 [508.7 to 1341.7] | 1288.0 [570.8 to 2906.4] | 1263.5 [794.7 to 2009.0] | 1149.0 [672.9 to 1961.8]
  Day 28: number analyzed (Participants) | 25 | 19 | 26 | 26 | 23 | 27 | 25 | 28 | 21 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 28 | 1218.3 [609.8 to 2433.7] | 1233.2 [658.4 to 2309.7] | 1471.1 [841.2 to 2572.7] | 953.8 [549.5 to 1655.4] | 754.4 [464.2 to 1226.0] | 1198.8 [688.3 to 2088.0] | 1310.7 [797.3 to 2154.5] | 1246.3 [710.3 to 2187.0] | 1086.0 [619.5 to 1903.7] | 1491.7 [983.7 to 2262.0] | 1940.6 [1259.0 to 2991.2] | 8866.0 [6415.5 to 12252.6] | 13710.2 [10111.0 to 18590.5] | 10202.3 [6715.1 to 15500.5] |  |  |  |  |  |
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 29 | 39 | 14 | 35 | 42
  Day 29 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 10170.0 [7301.6 to 14165.2] | 1172.6 [630.4 to 2181.1] | 818.6 [510.4 to 1313.0] | 1251.3 [563.1 to 2780.5] | 9284.7 [6772.0 to 12729.9] | 8508.2 [5798.6 to 12484.1]
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 36 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 5938.0 [3771.8 to 9348.2] | 4248.1 [2787.2 to 6474.8] | 8348.3 [5370.9 to 12976.3] | 9415.5 [7120.6 to 12450.1] | 8518.7 [5970.1 to 12155.2]
  Day 56: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 56 | 5051.3 [3144.0 to 8115.7] | 8644.5 [6368.1 to 11734.7] | 5651.7 [4159.3 to 7679.4] | 3909.2 [2620.5 to 5831.7] | 6655.7 [4670.1 to 9485.5] | 7585.7 [5687.6 to 10117.3] | 3296.3 [2075.7 to 5234.7] | 9110.9 [5865.5 to 14152.2] | 4762.7 [2918.8 to 7771.4] | 10733.0 [7902.0 to 14578.1] | 9544.8 [6846.7 to 13306.1] | 7083.6 [5125.3 to 9790.1] | 10333.3 [7485.5 to 14264.4] | 7801.7 [5379.1 to 11315.4] |  |  |  |  |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 57 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 9761.9 [6487.9 to 14688.1] | 5961.1 [4365.7 to 8139.7] | 8689.8 [6309.5 to 11968.1] | 7673.7 [5733.9 to 10269.7] | 7610.5 [5336.3 to 10854.0]
  Day 208: number analyzed (Participants) | 25 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 28 | 19 | 25 | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
  Day 208 | 2805.0 [1665.3 to 4724.8] | 3797.7 [2654.3 to 5433.8] | 2757.9 [1631.0 to 4663.4] | 2575.3 [1695.6 to 3911.3] | 2861.7 [2000.7 to 4093.2] | 3086.6 [2194.7 to 4341.0] | 2239.3 [1451.7 to 3454.4] | 4668.9 [3069.6 to 7101.4] | 2349.9 [1405.2 to 3929.8] | 4661.9 [3401.9 to 6388.5] | 4450.1 [2994.6 to 6613.0] | 4004.2 [2834.4 to 5656.7] | 4807.4 [3225.4 to 7165.3] | 4177.3 [2914.0 to 5988.2] |  |  |  |  |  |
  Day 211: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 39 | 14 | 35 | 42
  Day 211 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 5710.0 [3654.0 to 8922.7] | 3949.0 [2991.2 to 5213.6] | 4825.8 [3063.2 to 7602.6] | 5389.0 [4070.1 to 7135.2] | 5415.4 [3633.4 to 8071.3]
  Year 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 26 | 37 | 10 | 32 | 35
  Year 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1513.3 [897.0 to 2553.2] | 2344.8 [1508.6 to 3644.5] | 1465.5 [1039.9 to 2065.3] | 4160.4 [1968.6 to 8792.4] | 2244.0 [1462.9 to 3442.1] | 2380.4 [1507.4 to 3759.2]
  Year 3: number analyzed (Participants) | 24 | 19 | 27 | 26 | 23 | 27 | 25 | 28 | 22 | 27 | 19 | 25 | 24 | 24 | 21 | 24 | 35 | 13 | 29 | 37
  Year 3 | 1643.9 [850.8 to 3176.6] | 1874.7 [1066.5 to 3295.6] | 1756.7 [1193.6 to 2585.3] | 1159.4 [731.0 to 1838.7] | 1193.5 [780.4 to 1825.4] | 1385.2 [946.0 to 2028.2] | 1425.3 [844.2 to 2406.6] | 1705.3 [1024.2 to 2839.3] | 1166.5 [608.1 to 2237.6] | 1775.4 [1208.6 to 2608.1] | 1783.7 [1093.8 to 2909.0] | 1880.8 [1254.3 to 2820.4] | 2079.5 [1465.2 to 2951.4] | 1946.0 [1303.7 to 2904.8] | 1202.9 [682.0 to 2121.6] | 2200.3 [1284.6 to 3768.8] | 1771.1 [1276.4 to 2457.6] | 2155.0 [1293.4 to 3590.8] | 2297.5 [1422.8 to 3709.9] | 2304.2 [1369.0 to 3878.4]
  Year 4: number analyzed (Participants) | 23 | 19 | 26 | 26 | 23 | 26 | 23 | 28 | 22 | 28 | 19 | 25 | 23 | 24 | 20 | 18 | 22 | 11 | 20 | 27
  Year 4 | 1580.2 [856.2 to 2916.6] | 2128.6 [1214.1 to 3732.0] | 1828.6 [1183.6 to 2825.2] | 1234.2 [791.8 to 1923.6] | 1283.8 [870.2 to 1894.0] | 1714.5 [1133.1 to 2594.2] | 2114.3 [1369.8 to 3263.4] | 1858.2 [1107.6 to 3117.5] | 1115.2 [597.5 to 2081.7] | 1762.5 [1170.1 to 2655.0] | 2173.9 [1287.5 to 3670.6] | 1702.1 [976.9 to 2965.5] | 2766.1 [1630.1 to 4694.0] | 2044.1 [1416.3 to 2950.2] | 1254.0 [743.5 to 2115.0] | 1514.3 [895.9 to 2559.5] | 1267.2 [788.9 to 2035.5] | 1806.5 [1032.7 to 3160.1] | 2466.9 [1489.0 to 4086.9] | 1823.5 [1089.5 to 3052.0]
  Year 5: number analyzed (Participants) | 21 | 19 | 26 | 24 | 23 | 26 | 24 | 27 | 22 | 25 | 19 | 24 | 21 | 24 | 19 | 8 | 15 | 10 | 10 | 17
  Year 5 | 1159.9 [587.5 to 2289.8] | 2232.6 [1270.8 to 3922.1] | 1702.6 [1091.4 to 2656.0] | 1135.0 [709.5 to 1815.7] | 1177.1 [774.7 to 1788.5] | 1545.6 [952.6 to 2507.9] | 1410.6 [927.5 to 2145.5] | 2047.9 [1097.6 to 3821.1] | 1265.5 [682.2 to 2347.3] | 2037.4 [1364.0 to 3043.1] | 1648.1 [989.0 to 2746.2] | 1746.6 [1149.0 to 2655.0] | 2225.0 [1305.9 to 3791.0] | 1624.0 [1073.2 to 2457.7] | 1241.5 [726.4 to 2121.8] | 1076.0 [406.2 to 2850.3] | 912.7 [529.7 to 1572.6] | 1187.7 [680.8 to 2071.8] | 1522.7 [936.1 to 2476.8] | 2097.3 [1285.7 to 3421.1]

ADVERSE EVENTS:
Time Frame: From the time of informed consent signed in this extension study up to end of study (approximately 5 years when combined with the NOR-107, 210 and 204)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose: Eligible participants who received Hepatitis A vaccine, IM, on Day 1, followed by norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MLP and 500 µg aluminium hydroxide, IM, on Day 28 in previous study NOR-107 were enrolled at 3rd year post-primary vaccination in this study.
Arm/Group | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose | NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose | NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/19 | 0/27 | 0/27 | 0/23 | 0/27 | 0/25 | 0/28 | 0/22 | 0/28 | 0/21 | 0/25 | 0/24 | 0/24 | 0/24 | 1/29 | 3/39 | 0/14 | 2/35 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/19 | 1/27 | 1/27 | 0/23 | 0/27 | 0/25 | 0/28 | 0/22 | 0/28 | 0/21 | 0/25 | 0/24 | 0/24 | 1/24 | 2/29 | 5/39 | 0/14 | 2/35 | 2/42
Other Adverse Events (participants affected / at risk) | 0/25 | 0/19 | 0/27 | 0/27 | 0/23 | 0/27 | 0/25 | 0/28 | 0/22 | 0/28 | 0/21 | 0/25 | 0/24 | 0/24 | 0/24 | 0/29 | 0/39 | 0/14 | 0/35 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 50 μg,1-Dose (N=25) | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 50 μg,1-Dose (N=19) | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 50 μg,1-Dose (N=27) | NOR-107: GI.1/GII.4 (15/15/500) μg- MPL 15 μg,1-Dose (N=27) | NOR-107: GI.1/GII.4 (15/50/500) μg- MPL 15 μg,1-Dose (N=23) | NOR-107: GI.1/GII.4 (50/50/500) μg- MPL 15 μg,1-Dose (N=27) | NOR-107: GI.1/GII.4 (15/15/500) μg,1-Dose (N=25) | NOR-107: GI.1/GII.4 (15/50/500) μg,1-Dose (N=28) | NOR-107: GI.1/GII.4 (50/50/500) μg,1-Dose (N=22) | NOR-107: GI.1/GII.4 (50/150/500) μg,1-Dose (N=28) | NOR-107: GI.1/GII.4 (15/50/167) μg,1-Dose (N=21) | NOR-107: GI.1/GII.4 (15/50/500) μg,2-Dose (N=25) | NOR-107: GI.1/GII.4 (50/150/500) μg,2-Dose (N=24) | NOR-107: GI.1/GII.4 (15/50/167) μg,2-Dose (N=24) | NOR-210: GI.1/GII.4 (15/50/500) µg, 1-Dose (N=24) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 1-Dose (N=29) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 60-94 Yrs) (N=39) | NOR-204: GI.1/GII.4 (15/50/500) µg, 1-Dose (Age: 18-49 Yrs) (N=14) | NOR-204: GI.1/GII.4 (15/50/500) µg - MPL 15 µg, 2-Dose (N=35) | NOR-204: GI.1/GII.4 (15/50/500) µg, 2-Dose (N=42)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Episcleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurodegenerative disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT03039790/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT03039790/SAP_001.pdf